CLINICAL TRIAL: NCT06380686
Title: Head and Neck Carcinoma Clinical Research Platform for Molecular and Blood-based
Brief Title: Head and Neck Carcinoma Clinical Research Platform for Molecular and Blood-based Biomarkers, Treatment and Outcome
Acronym: HEAT
Status: Recruiting | Type: Observational
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AIO-KHT-0322/ass
Record Dates: First submitted 2024-04-12; First posted 2024-04-24 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity; Squamous Cell Carcinoma of the Oropharynx; Squamous Cell Carcinoma of the Hypopharynx; Squamous Cell Carcinoma of the Larynx
Keywords: SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — For future translational research projects, the location of tissue samples in local pathologies will be recorded for patients who have consented to the use of their tissue samples, creating a decentralized biobank.
  Future translational research projects cannot be pre-defined. Any future translational research project will be described in detail in a project plan and submitted to an ethics committee for review and approval.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — Demography, Social history, Riskfactors, Relevant medical history, Oncological family history, Disease & treatment history, Molecular Pathology and Results, Treatment data, Response data, progession free survial, overall survival.

SUMMARY:
Prospective, open, non-interventional, multi-center clinical registry study with the aim to establish a comprehensive research platform reflecting the real-world treatment landscape for recurrent/metastatic head and neck tumor patients.

DETAILED DESCRIPTION:
The advent of checkpoint inhibitors has changed the treatment landscape in SCCHN and new treatment sequences have entered clinical practice.

More in-depth knowledge of tumor biomarkers are important measures for optimization of treatment strategies in SCCHN. In addition to this, investigations may involve other assessments, which will be explored separately, such as molecular testing. These tests are then linked to the core data set and will allow to associate such measures with outcomes. This concept is flexible and allows for rapid integration of contemporary research questions in a timely manner.

Furthermore, insights into the treatment reality for recurrent/metastatic salivary gland carcinoma and other rare tumor entities (SNUC, etc.) are urgently needed, as there is currently no established standard of care.

The monoclonal antibody cetuximab in combination with platinum and fluorouracil (EXTREME) has been the standard of care for recurrent or metastatic (r/m) SCCHN for over a decade.1 Recently, the immune checkpoint inhibitors (CPIs) nivolumab and pembrolizumab have changed the therapeutic landscape of patients with r/m SCCHN. Nivolumab is considered as therapeutic standard after failure of platinum-based therapy based on the results of the phase III Checkmate-141 trial.2 In addition, pembrolizumab has become the new standard in the first-line setting in combination with platinum/fluorouracil chemotherapy or as monotherapy for patients with programmed cell death ligand 1 (PD-L1) positive tumors based on the data from the phase III Keynote-048 trial.3 Moreover, cetuximab in combination with platinum and docetaxel (TPEx) has emerged as a less toxic alternative to the EXTREME regimen.4 Due to the shifting first-line treatment landscape, data to guide contemporary 2nd line therapy are scarce and the optimal treatment sequence remains vague.2,5,6 The implementation of biomarkers and selection of patients in a real-world setting are areas of academic interest. In addition, the assessment of treatment outcomes in rare entities are underrepresented in pivotal trials, and as a matter of fact, may be completely excluded. However, broad labels permit the use of novel agents, but a larger body of evidence is needed to substantiate such treatment choices. HEAT seeks to address these questions by inclusion of a real-world patient population and continuous assessment of oncological outcomes by means of a core clinical data set implemented into HEAT.

Overall, HEAT is a study platform, which continuously assesses clinical outcomes and modularly integrates additional measures to enable rapid answers to research questions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to understand and willing to sign written informed consent
* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck (oral cavity, oropharynx, hypopharynx or larynx)
* Patients not amenable for curative treatment who receive palliative systemic treatment or best supportive care
* Informed consent no later than four weeks after start of first-line palliative systemic treatment. For patients receiving "best supportive care only": no later than six weeks after diagnosis/recurrence or metastatic disease

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically or cytologically confirmed malignancy of the head neck area including but not limited to
  * squamous cell carcinoma (SCC) of the oral cavity, oropharynx, hypopharynx or larynx
  * not amenable for curative treatment who receive palliative systemic treatment or best supportive care.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic factors | 3 years
  Highest level of education, Employment status, Current professional activity, Professional risk factors, Level of self-sufficiency, Care degree
Treatments | 3 years
  Types of local therapies (surgery, radiotherapy, radiochemotherapy), systemic therapy and therapeutic sequences
Response rates | 3 years
  Response rates
Treatment decision | 3 years
  Physician-reported parameters affecting treatment decision
Progression-free survival | 3 years
  Progression-free survival
Time-to-treatment-failure | 3 years
  Time-to-treatment-failure
Overall survival | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Victor Grünwald, Prof. Dr., Study Director — Universitätsklinikum Essen; Michael Pogorzelski, Dr., Principal Investigator — Universitätsklinikum Essen
Locations (2):
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Onkologie/Studienzentrum am Raschplatz GbR, Hanover

IPD SHARING:
Plan to Share IPD: No